CLINICAL TRIAL: NCT05773053
Title: A Prospective, Double-blind, Randomized, Placebo-controlled, Multicenter Study to Investigate the Efficacy and Safety of NT 201 Doses in the Treatment of Platysma Prominence
Brief Title: A Study of NT 201 Doses in the Treatment of Platysma Prominence
Acronym: PAOLA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merz Aesthetics GmbH (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M602011078
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Platysma Prominence
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NT 201 Dose 1 (Experimental): Subjects will receive Dose 1.
  Interventions: Drug: NT 201
- NT 201 Dose 2 (Experimental): Subjects will receive Dose 2.
  Interventions: Drug: NT 201
- NT 201 Dose 3 (Experimental): Subjects will receive Dose 3.
  Interventions: Drug: NT 201
- Placebo (Placebo Comparator): Subjects will receive matching placebo.
  Interventions: Drug: NT 201 Placebo

INTERVENTIONS:
Drug: NT 201 — Clostridium botulinum neurotoxin type A (150 kiloDalton [kD], free of complexing proteins) powder for solution for injection.
  Other Names: IncobotulinumtoxinA; Xeomin/Bocouture; Xeomin Cosmetic; Xeomeen
  Arms: NT 201 Dose 1; NT 201 Dose 2; NT 201 Dose 3
Drug: NT 201 Placebo — NT 201 Matching-placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of NT 201 in adults with moderate to severe platysma prominence.

ELIGIBILITY:
Inclusion Criteria:

* Presence of four (medial and lateral, left and right) prominent platysmal bands
* Moderate to severe platysmal bands as assessed by the investigator and subject on the MAPS-D at maximum contraction

Exclusion Criteria:

* Any serious disease or disorder (medical or psychiatric) that could interfere with the safe completion of treatment or compromise subject safety
* Botulinum toxin treatment in the face (below the lower orbital rim), neck, or chest within the last 12 months prior to study treatment
* History of lower face surgery, neck or chest surgery, aesthetic procedures (e.g., ablative skin resurfacing, laser, chemical peel, micro-focused ultrasound, deoxycholic acid injections, micro-needling, non-surgical fat reduction procedure), and orthodontic procedures (e.g., braces) in the 12 months prior to study treatment
* Previous use of any permanent (non-biodegradable) or semi-permanent (e.g., calcium hydroxylapatite, poly-L-lactic acid, polymethyl methacrylate, etc.) facial tissue augmentation therapy, lifting sutures, permanent implants or autologous fat to the lower face (i.e., below the level of the bottom of the nose), neck, or chest within 24 months prior to study treatment
* Previous use of any hyaluronic acid based or collagen based biodegradable facial tissue augmentation therapy to the lower face (i.e., below the level of the bottom of the nose), neck, or chest within 12 months prior to study treatment
* Any medical condition that may put the subject at increased risk with exposure to botulinum toxin of any serotype, including myasthenia gravis, Lambert-Eaton-Syndrome, amyotrophic lateral sclerosis, or any other disorder that might interfere with neuromuscular function
* Female of childbearing potential not using a highly effective method of birth control, planning to get pregnant, or pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Change From Baseline on the MAPS-D Score at Maximum Contraction as Assessed by the Investigator at Visit 4 (V4) | Baseline (Screening Visit), Week 2 (V4)
  The platysma area will be assessed live by the investigator at maximum contraction and graded according to the validated five-point Merz Aesthetic Platysma Scale-Dynamic (MAPS-D). Scores range from Grade 1 (none to minimal) to Grade 5 (very severe).

SECONDARY OUTCOMES:
Change From Baseline on the MAPS-D Score at Maximum Contraction as Assessed by the Subject at V4 | Baseline (Screening Visit), Week 2 (V4)
  The platysma area will be assessed by the subjects at maximum contraction and graded according to the validated five-point MAPS-D. Scores range from Grade 1 (none to minimal) to Grade 5 (very severe).
Number of Subjects With Related Treatment Emergent Adverse Events (Related TEAEs) | Baseline up to Week 17/End of Study
  TEAEs are defined as adverse events (AEs) with onset or worsening on or after date and time of first dose of study treatment. An AE is considered to be related if a causal relationship between NT 201 and the AE is at least reasonably possible.

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (7):
- United States (7):
  - Merz Investigation Site #0010170, Washington D.C., District of Columbia
  - Merz Investigational Site #0010453, Aventura, Florida
  - Merz Investigation Site #0010470, Coral Gables, Florida
  - Merz Investigation Site #0010105, Metairie, Louisiana
  - Merz Investigation Site #0010471, Verona, New Jersey
  - Merz Investigation Site #0010469, New York, New York
  - Merz Investigation Site #0010405, New York, New York

IPD SHARING:
Plan to Share IPD: No